CLINICAL TRIAL: NCT05033249
Title: The Utility of Immature Granulocyte Count and Percentage on the Prediction of Acute Appendicitis in the Suspected Acute Appendicitis According to the ALVARADO Scoring System: A Retrospective Cohort Study
Brief Title: The Utility of Immature Granulocyte Count on the Prediction of Acute Appendicitis in the Suspected Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Özlem Güler (Unknown); Filiz Alkan Baylan (Unknown)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Other Study IDs: 181
Record Dates: First submitted 2021-06-19; First posted 2021-09-02 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Appendicitis
Keywords: Acute appendicitis; Computed Tomography; Immature granulocyte count; Immature granulocyte percentage; Alvarado Scoring System
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: Alvarado Score 4 - 7 Normal according to the initial computed tomographic evaluation
  Interventions: Diagnostic Test: Immature granulocyte count; Diagnostic Test: Immature granulocyte percentage
- Patient: Alvarado Score 4 - 7 Acute appendicitis according to the initial computed tomographic evaluation
  Interventions: Diagnostic Test: Immature granulocyte count; Diagnostic Test: Immature granulocyte percentage

INTERVENTIONS:
Diagnostic Test: Immature granulocyte count — Automatically calculated immature granulocyte count in white blood cell count
Diagnostic Test: Immature granulocyte percentage — Automatically calculated immature granulocyte percentage in white blood cell count

SUMMARY:
Acute appendicitis is the most common cause of abdominal pain requiring surgery in the emergency department. The whole life acute appendicitis rate is 7%. Only half of the patients with acute appendicitis are presented with typical periumbilical pain following by nausea, vomiting, and the migration of pain to the right lower quadrant. The diagnosis of acute appendicitis is based on the patient's medical history, physical examination, and laboratory findings. The Alvarado scoring system (ASS), recommends discharge, observation, and surgical intervention to patients. However, such scoring systems should not be used as the only method in diagnosis. Increased imaging use in patients with suspected acute appendicitis improved the rate of correct diagnosis. American College of Radiology Appropriateness Criteria (ACR) recommends computerized tomography (CT) as the primary imaging method to confirm the diagnosis of acute appendicitis in adults. However, CT imaging has some disadvantages, such as radiation exposure, undesirable effects associated with the use of contrast agents, and increased workload in the emergency room. The count of immature granulocytes (IGC), which is an indicator of increased activation of the bone marrow, and the percentage of IG (IGP), which is the ratio of IGs to the total white blood cell count, are also has been used differentiation of complicated acute appendicitis from uncomplicated acute appendicitis, and other inflammatory pathologies. Nowadays automatic blood analyzers can easily measure the amount and percentage of IGs simultaneously in a complete blood count test with advances in technology.

It is aimed to investigate the utility of IGC and IGP on the prediction of suspected acute appendicitis according to the ASS and its effect on the need for CT scanning.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of abdominal pain requiring surgery in the emergency department. The highest incidence of acute appendicitis is in the 2nd and 3rd decades of life, but it can be seen at any age. There is a 7% chance that a person will have appendicitis during life. Only half of the patients with acute appendicitis are presented with typical periumbilical pain following by nausea, vomiting, and the migration of pain to the right lower quadrant. The diagnosis of acute appendicitis is based on the patient's medical history, physical examination, and laboratory findings. Various clinical prediction rules have been developed to increase diagnostic accuracy. The most accepted among these is the Alvarado scoring system (ASS). ASS classifies patients as low, moderate, and high-risk groups for acute appendicitis. Accordingly, it recommends discharge, observation, and surgical intervention to patients. However, such scoring systems should not be used as the only method in diagnosis.

Increased imaging use in patients with suspected acute appendicitis improved the rate of correct diagnosis. American College of Radiology Appropriateness Criteria (ACR) recommends computerized tomography (CT) as the primary imaging method to confirm the diagnosis of acute appendicitis in adults. However, CT imaging has some disadvantages, such as radiation exposure, undesirable effects associated with the use of contrast agents, and increased workload in the emergency room.

Numerous inflammatory parameters adapted from complete blood count parameters can be used in infectious inflammatory processes such as acute appendicitis, pyelonephritis, and non-infectious conditions such as differentiation of tumoral masses from benign lesions, and determining survival in acute myocardial infarction. Among these parameters, neutrophil-lymphocyte ratio, platelet lymphocyte ratio, and lymphocyte monocyte ratio were used in previous studies. Similarly, the number of immature granulocytes (IGC), which is an indicator of increased activation of the bone marrow, and the percentage of IG (IGP), which is the ratio of IGs to the total white blood cell count, are also has been used in acute necrotizing pancreatitis, differentiation of complicated acute appendicitis from uncomplicated acute appendicitis, pyelonephritis, sepsis, thyroid gland malignancies, and renal cell carcinomas. Previously the determination of the number of IGs could be possible based on counting granulocyte precursor cells during the direct microscopic examination. Nowadays automatic blood analyzers can easily measure the amount and percentage of IGs simultaneously in a complete blood count test with advances in technology. Immature granulocyte (IG) in peripheral blood is an indicator of increased bone marrow activity. It has been reported in previous studies that IGC and IGP increase in infection and sepsis, and are more reliable markers in the diagnosis of acute appendicitis than other hematological parameters.

This study aimed to investigate the utility of IGC and IGP on the prediction of suspected acute appendicitis according to the ASS and its effect on the need for CT scanning.

MATERIALS AND METHODS Study design and setting This study is a retrospective cohort analysis involving adult patients who were admitted to the emergency department of a university hospital between January 2019 and July 2019 due to abdominal pain and suspected acute appendicitis according to ASS. Local ethics committee approval was received for the study (ethics committee approval number 2019/11/06). Because the study design is retrospective, the signed informed consent of patients is not required. All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Declaration of Helsinki and its later amendments or comparable ethical standards.

Patient Selection and Data Collection Adult patients who admitted to the Emergency Department of Kahramanmaras Sutcu Imam University hospital due to abdominal pain and had an ASS between 4-7, and whose initial imaging technique was CT were included in the study. ASS scores of the patients were calculated retrospectively by examining patients' medical records. Patients were used other imaging methods, underwent surgery without imaging, followed by medical treatment without surgery, pregnant, under the age of 18, with incomplete medical records, and with additional diseases (such as underlying hematologic or rheumatologic disease, other concurrent infectious diseases) and treated with granulocyte colony-stimulating factors, glucocorticoids, or other immunosuppressants that may affect inflammation markers were excluded from the study.

Electronic files of the patients recorded in the hospital database were reviewed by the investigators. Demographic data (age, gender), laboratory values, tomography reports, and pathological diagnoses were recorded. The diagnosis was also confirmed histopathologically in all patients diagnosed with acute appendicitis according to the result of tomography.

The white blood cell count (WBC), neutrophil count, lymphocyte count, IGC, and IGP were obtained from the blood sample taken at the time of the patient's first admission to the hospital using the Sysmex XN-3000 (Sysmex Corporation, Kobe, Japan) device. Neutrophil/lymphocyte ratio (NLR) was calculated manually from hemogram results. The patients were divided into two groups as those with acute appendicitis (appendicitis positive group, Group-P) and non-appendicitis (appendicitis negative group, Group-N) according to the result of tomography.

Statistical analysis The data were analyzed with the IBM Statistical Package for the Social Sciences (SPSS ver. 20) program. The compliance of continuous variables to normal distribution was evaluated with the Shapiro-Wilk test. An independent sample t-test was used to compare the data that complied with the normal distribution and the Mann Whitney-U test was used for those that did not comply with the normal distribution. Pearson test was used for correlation analysis of normally distributed parameters, and the Spearman test was used for correlation analysis of non-normally distributed parameters. Multivariate analysis was performed with parameters found to be significant in the evaluation of univariate analysis and predictive values of preoperative blood parameters were calculated. The Chi-square test was used to analyze categorical variables. p<0.05 value was considered significant. The Receiver Operating Characteristic (ROC) curve analysis was used to evaluate the success of laboratory parameters in predicting acute appendicitis diagnosis. The area under the curve (AUC), sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy rate were calculated for parameters with a statistically significant difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients complaining about abdominal pain
* Calculated ALVARADO Score 4-7
* Whose initial imaging technique was CT

Exclusion Criteria:

* Patients diagnosed with other imaging methods (eg, ultrasonography)
* Patients who underwent surgery without imaging modalities
* Patients who were followed by medical treatment without surgery
* Pregnant patients
* Age <18
* Patients with incomplete medical records
* Patients with additional diseases which can affect the blood parameters (such as underlying hematologic or rheumatologic disease, laignancies, other concurrent infectious diseases)
* Patients whom were treated with granulocyte colony-stimulating factors, glucocorticoids, or other immunosuppressants that may affect inflammation markers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal pain admitted to the emergency room and whose calculated ALVARADO score was between 4 and 7. According to this result computed tomographic evaluation applied to these patients.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The utility of Immature granulocyte count on determining clinically suspected acute appendicitis cases and diminishing computed tomography need | January 2019 - July 2019
  Automatically counted immature granulocyte count can help to determine acute appendicitis cases and diminish the need for computed tomography in patients who admitted to the emergency room and ALVARADO score between 4 - 7.
The utility of Immature granulocyte percentage on determining clinically suspected acute appendicitis cases and diminishing computed tomography need | January 2019 - July 2019
  Automatically calculated immature granulocyte percentage can help to determine acute appendicitis cases and diminish the need for computed tomography in patients who admitted to the emergency room and ALVARADO score between 4 - 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohle R, O'Reilly F, O'Brien KK, Fahey T, Dimitrov BD. The Alvarado score for predicting acute appendicitis: a systematic review. BMC Med. 2011 Dec 28;9:139. doi: 10.1186/1741-7015-9-139. PMID 22204638
- [Background] Hosseini M, Tizmaghz A, Shabestanipour G, Aein A, Otaghvar H. The Frequency of Different Clinical Presentation of Appendicitis, Complications and Prognosis in Elderly. Annu Res Rev Biol. 2014;4(24):4381-8
- [Background] Shuaib A, Shuaib A, Fakhra Z, Marafi B, Alsharaf K, Behbehani A. Evaluation of modified Alvarado scoring system and RIPASA scoring system as diagnostic tools of acute appendicitis. World J Emerg Med. 2017;8(4):276-280. doi: 10.5847/wjem.j.1920-8642.2017.04.005. PMID 29123605
- [Background] Dal F, Cicek Y, Pekmezci S, Kocazeybek B, Tokman HB, Konukoglu D, Simsek O, Taner Z, Sirekbasan S, Uludag SS. Role of Alvarado score and biological indicators of C-reactive protein, procalicitonin and neopterin in diagnosis of acute appendicitis. Ulus Travma Acil Cerrahi Derg. 2019 May;25(3):229-237. doi: 10.5505/tjtes.2018.57362. PMID 31135946
- [Background] Tintinalli JE, Stapczynski JS, Ma OJ, Cline DM, Cydulka Rk MG, editor. Gastrointestinal Emergencies. In: Tintinalli's Emergency Medicine: A Comprehensive Study Guide. 7th ed. New York: McGraw-Hill Medical; 2010
- [Background] Rosen MP, Ding A, Blake MA, Baker ME, Cash BD, Fidler JL, Grant TH, Greene FL, Jones B, Katz DS, Lalani T, Miller FH, Small WC, Spottswood S, Sudakoff GS, Tulchinsky M, Warshauer DM, Yee J, Coley BD. ACR Appropriateness Criteria(R) right lower quadrant pain--suspected appendicitis. J Am Coll Radiol. 2011 Nov;8(11):749-55. doi: 10.1016/j.jacr.2011.07.010. PMID 22051456
- [Background] Smith MP, Katz DS, Lalani T, Carucci LR, Cash BD, Kim DH, Piorkowski RJ, Small WC, Spottswood SE, Tulchinsky M, Yaghmai V, Yee J, Rosen MP. ACR Appropriateness Criteria(R) Right Lower Quadrant Pain--Suspected Appendicitis. Ultrasound Q. 2015 Jun;31(2):85-91. doi: 10.1097/RUQ.0000000000000118. PMID 25364964
- [Background] Unal Y, Barlas AM. Role of increased immature granulocyte percentage in the early prediction of acute necrotizing pancreatitis. Ulus Travma Acil Cerrahi Derg. 2019 Mar;25(2):177-182. doi: 10.14744/tjtes.2019.70679. PMID 30892679
- [Background] Unal Y. A new and early marker in the diagnosis of acute complicated appendicitis: immature granulocytes. Ulus Travma Acil Cerrahi Derg. 2018 Sep;24(5):434-439. doi: 10.5505/tjtes.2018.91661. PMID 30394497
- [Background] Bozan MB, Yazar FM, Kale IT, Yuzbasioglu MF, Boran OF, Azak Bozan A. Delta Neutrophil Index and Neutrophil-to-Lymphocyte Ratio in the Differentiation of Thyroid Malignancy and Nodular Goiter. World J Surg. 2021 Feb;45(2):507-514. doi: 10.1007/s00268-020-05822-6. Epub 2020 Oct 16. PMID 33067685
- [Background] Barut O, Demirkol MK, Bilecan EB, Sahinkanat T, Resim S. The Delta Neutrophil Index is an Early Predictive Marker of Acute Pyelonephritis in Patients with Ureteral Stone. J Coll Physicians Surg Pak. 2020 Nov;30(11):1149-1154. doi: 10.29271/jcpsp.2020.11.1149. PMID 33222730
- [Background] Kong T, Park YS, Lee HS, Kim S, Lee JW, You JS, Chung HS, Park I, Chung SP. The delta neutrophil index predicts development of multiple organ dysfunction syndrome and 30-day mortality in trauma patients admitted to an intensive care unit: a retrospective analysis. Sci Rep. 2018 Nov 30;8(1):17515. doi: 10.1038/s41598-018-35796-4. PMID 30504778
- [Background] Shin DH, Cho YS, Cho GC, Ahn HC, Park SM, Lim SW, Oh YT, Cho JW, Park SO, Lee YH. Delta neutrophil index as an early predictor of acute appendicitis and acute complicated appendicitis in adults. World J Emerg Surg. 2017 Jul 24;12:32. doi: 10.1186/s13017-017-0140-7. eCollection 2017. PMID 28747992
- [Background] Barut O, Demirkol MK, Kucukdurmaz F, Sahinkanat T, Resim S. Pre-treatment Delta Neutrophil Index as a Predictive Factor in Renal Cell Carcinoma. J Coll Physicians Surg Pak. 2021 Feb;31(2):156-161. doi: 10.29271/jcpsp.2021.02.156. PMID 33645181